CLINICAL TRIAL: NCT00078897
Title: Phase III Study of the Effects of Selenium on Adenomatous Polyp Recurrence
Brief Title: Selenium for Prevention of Adenomatous Colorectal Polyps
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Concluded - Terminated by PI
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDR0000353185; P30CA023074 (NIH); P01CA041108 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer; Adenomatous Colorectal Polyps; Precancerous Condition
Keywords: colon cancer; rectal cancer; colorectal cancer; adenomatous polyp
MeSH Terms: conditions — Colorectal Neoplasms; Precancerous Conditions; Colonic Neoplasms; Rectal Neoplasms; Adenomatous Polyps | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selenium (Active Comparator): Participants receive oral selenium 200 mcg once daily.
  Interventions: Drug: Selenium
- Placebo (Placebo Comparator): Participants receive oral placebo once daily.
  Interventions: Drug: Selenium

INTERVENTIONS:
Drug: Selenium — Participants will be randomized either to selenium or placebo, taking the randomized intervention for 3 to 5 years, depending on when their recommended follow up colonoscopy is scheduled.
  Other Names: SelenoExcell

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Selenium may be effective in preventing the recurrence of adenomatous colorectal polyps.

PURPOSE: This randomized phase III trial is studying selenium to see how well it works in preventing the recurrence of polyps in patients with adenomatous colorectal polyps.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effects of selenium vs placebo on the recurrence of adenomatous colorectal polyps, in terms of histologic type, degree of dysplasia, number, size, and location, in patients with adenomatous colorectal polyps.
* Compare the type, incidence, and outcome of side effects in patients treated with these regimens.
* Determine patient adherence to long-term treatment with these regimens.

Secondary

* Determine the effects of regimen modification by baseline blood selenium level, low-dose aspirin, selenoprotein genetic marker polymorphisms (e.g., GPx-1, GPx-2, and SEP15)
* Determine the effects of low-dose aspirin (81 mg/day) modification by ornithine decarboxylase promoter genotype, and toxicity by slow-metabolizer genotypes of the cytochrome p450 2C9 and UT1A6 loci in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to use of low-dose (≤ 81 mg/day) aspirin (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral selenium once daily.
* Arm II: Patients receive oral placebo once daily. In both arms, treatment continues for up to 5 years* in the absence of disease progression or unacceptable toxicity.

Patients undergo follow-up colonoscopy approximately 5 years* after baseline colonoscopy.

NOTE: Some patients will continue participation for up to 7 and a half years

PROJECTED ACCRUAL: A total of 1,600 patients with an adenoma will be randomized to this study, followed by a second group of randomization of 200 patients with at least one advanced adenoma (at baseline) for a substudy. Total planned randomizations = 1,800 participants.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenomatous polyps
* Meets the following criteria by colonoscopy (performed within the past 6 months):

  * Cecum was totally visualized or reached
  * At least 90% visualization of colon surface area
  * Removed at least 1 adenomatous polyp of at least 3 mm in size during procedure (For the Advanced Adenoma Sub-study: Removal of at least 1 advanced colorectal adenomatous polyp during procedure. An adenoma is considered advanced if it is 10 mm or greater in size, and/or has villous histology and/or shows high grade dysplasia)
  * Removed no more than 10 adenomatous polyps of any size by endoscopy
  * All other neoplastic and non-neoplastic colon polyps must have been completely removed (except for diminutive [less than 3 mm] sessile rectal polyps)
  * For the sub-study, at least 1 advanced adenomatous polyp defined as 10 mm or greater in size and/or has villous histology and/or shows high grade dysplasia
* No prior diagnosis of any of the following:

  * Colorectal cancer
  * Familial adenomatous polyposis
  * Ulcerative colitis
  * Crohn's disease
  * Hereditary non-polyposis colon cancer (HNPCC), defined as:

    * Histologically confirmed colorectal cancer in at least 3 relatives, 1 of whom is a first-degree relative of the other 2
    * Disease occurrence in at least 2 consecutive generations
    * Colorectal cancer diagnosis in at least 1 family member who is less than 50 years of age

      * Patients with a family history of colorectal cancer but who are not diagnosed with HNPCC are allowed
* No more than 1 prior segmental colon resection

PATIENT CHARACTERISTICS:

Age

* 40 to 80

Performance status

* SWOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin > 11 g/dL
* WBC 3,000 - 11,000/mm^3

Hepatic

* AST and ALT < 2 times upper limit of normal
* Bilirubin < 2.0 mg/dL

Renal

* Creatinine < 1.9 mg/dL

Cardiovascular

* No unstable* cardiac disease despite medication (e.g., diuretics or digitalis)
* No uncontrolled hypertension (i.e., systolic blood pressure ≥ 170 mm Hg and/or diastolic blood pressure ≥ 110 mm Hg) despite medication NOTE: *Unstable defined as unable to walk across the room without chest pain or shortness of breath

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception for at least 2 months before and during study treatment
* Resident of a clinical center metropolitan area or obtaining regular health care in a clinical metropolitan area for at least 6 months out of the year
* Must be able to swallow pills
* No unexpected weight loss of 10% or more within the past 6 months
* No prior rheumatoid arthritis
* No poorly controlled diabetes mellitus despite medication, defined as:

  * Blood sugar level ≥ 200 mg/dL on more than half of the readings taken within the past month
* No invasive malignancy within the past 5 years that required medical excision, radiotherapy, or chemotherapy except basal cell or squamous cell carcinoma

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent drugs that regulate the immune system

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* Prior enrollment in another adenoma prevention study allowed
* Concurrent routine aspirin (≤ 81 mg/day) allowed
* No regular use of non-steroidal anti-inflammatory drugs (NSAIDs)
* No concurrent enrollment in another research study using pharmacological cancer drugs, a cyclo-oxygenase-2 inhibitor, or selenium
* No other concurrent selenium unless dosage is ≤ 50 µg/day

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1621 (Actual)
Dates: Start 2005-01-20 (Actual); Primary Completion 2014-01-07 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Peter Lance, MD, Principal Investigator — University of Arizona
Locations (7):
- United States (7):
  - Veterans Affairs Medical Center - Phoenix, Phoenix, Arizona
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Cancer Center - Tucson Clinic, Tucson, Arizona
  - University of Colorado Cancer Center at UC Health Sciences Center, Denver, Colorado
  - Endoscopy Center of Western New York, Williamsville, New York
  - Baylor University Medical Center - Dallas, Dallas, Texas

REFERENCES:
- [Derived] Trejo MJ, Batai K, Chen Y, Brezina S, Chow HS, Ellis N, Lance P, Hsu CH, Pogreba-Brown K, Bishop M, Gsur A, Jacobs ET. Genome-Wide Association Study of Metachronous Colorectal Adenoma Risk among Participants in the Selenium Trial. Nutr Cancer. 2023;75(1):143-153. doi: 10.1080/01635581.2022.2096910. Epub 2022 Jul 9. PMID 35815403
- [Derived] Jacobs ET, Lance P, Mandarino LJ, Ellis NA, Chow HS, Foote J, Martinez JA, Hsu CP, Batai K, Saboda K, Thompson PA. Selenium supplementation and insulin resistance in a randomized, clinical trial. BMJ Open Diabetes Res Care. 2019 Feb 7;7(1):e000613. doi: 10.1136/bmjdrc-2018-000613. eCollection 2019. PMID 30899530
- [Derived] Thompson P, Roe DJ, Fales L, Buckmeier J, Wang F, Hamilton SR, Bhattacharyya A, Green S, Hsu CH, Chow HH, Ahnen DJ, Boland CR, Heigh RI, Fay DE, Martinez ME, Jacobs E, Ashbeck EL, Alberts DS, Lance P. Design and baseline characteristics of participants in a phase III randomized trial of celecoxib and selenium for colorectal adenoma prevention. Cancer Prev Res (Phila). 2012 Dec;5(12):1381-93. doi: 10.1158/1940-6207.CAPR-12-0204. Epub 2012 Oct 11. PMID 23060037
- [Derived] Solomon SD, Wittes J, Finn PV, Fowler R, Viner J, Bertagnolli MM, Arber N, Levin B, Meinert CL, Martin B, Pater JL, Goss PE, Lance P, Obara S, Chew EY, Kim J, Arndt G, Hawk E; Cross Trial Safety Assessment Group. Cardiovascular risk of celecoxib in 6 randomized placebo-controlled trials: the cross trial safety analysis. Circulation. 2008 Apr 22;117(16):2104-13. doi: 10.1161/CIRCULATIONAHA.108.764530. Epub 2008 Mar 31. PMID 18378608
- See also: Journal Article — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6272807/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through clinical centers in Arizona, Colorado, Texas, and New York following ambulatory colonoscopies. Eligible participants were between age 40 and 80 years and had undergone colonoscopic removal of one or more colorectal adenomas 3 mm or larger within six months prior to random assignment.
Period: Overall Study
Arm/Group | Selenium | Placebo
Started | 809 | 812
Completed | 685 | 689
Not Completed | 124 | 123

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selenium | Placebo | Total
Number analyzed (Participants) | 685 | 689 | 1374
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.9) | 63.1 (8.7) | 63.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 234 | 476
  Male | 443 | 455 | 898
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 39 | 64
  Not Hispanic or Latino | 660 | 650 | 1310
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 16 | 33
  White | 652 | 650 | 1302
  More than one race | 7 | 13 | 20
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 685 | 689 | 1374

OUTCOME MEASURES:

1. Primary Outcome: Number of Recurrent Adenomas at Surveillance Colonoscopy
Description: Detection of metachronous colorectal adenomas during follow-up, by treatment, in the original cohort. Surveillance colonoscopy is recommended 3 to 5 years after removal of colorectal adenoma(s). Participants will remain on the study intervention until their surveillance colonoscopy. Surveillance colonoscopy is determined by participants' GI physician.
Time Frame: 3 to 5 years after baseline colonoscopy
Measure: Number; unit: Adenomas
Arm/Group | Selenium | Placebo
Number analyzed (Participants) | 685 | 689
Adenomas | 302 | 295

2. Primary Outcome: Median Selenium Blood Levels at One Year.
Description: Adequate adherence to long-term selenium treatment as measured by blood selenium levels (ng/mL) at one year.
Time Frame: One year
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Selenium | Placebo
Number analyzed (Participants) | 685 | 689
ng/mL | 205.4 [100.7 to 367.6] | 140.0 [84.9 to 270.2]
Statistical Analysis 1: Comparison: Selenium; Test type: Other — Negative binomial regression; p = 0.68, Negative binomial regression; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.91 to 1.16]

ADVERSE EVENTS:
Arm/Group | Selenium | Placebo
All-Cause Mortality (participants affected / at risk) | 11/685 | 10/689
Serious Adverse Events (participants affected / at risk) | 228/685 | 226/689
Other Adverse Events (participants affected / at risk) | 0/685 | 0/689
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selenium (N=685) | Placebo (N=689)
Abdominal aortic aneurysm (Vascular disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 4
Acute appendicitis (Gastrointestinal disorders) | 1 | 3
Acute cholecystitis (Hepatobiliary disorders) | 0 | 3
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 48 | 67
Myocardial Infarction (Cardiac disorders) | 6 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 9
Allergic reaction (Immune system disorders) | 2 | 2
Angioedema (Immune system disorders) | 0 | 2
Angina (Cardiac disorders) | 12 | 12
Chest pain (Cardiac disorders) | 10 | 11
COPD (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Diverticulitis (Gastrointestinal disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Arthritis/Degenerative joint disease (Musculoskeletal and connective tissue disorders) | 18 | 16
Stroke/Transient ischemic attack (Nervous system disorders) | 10 | 10
Atrial fibrillation/arrhythmia (Cardiac disorders) | 13 | 9
Fracture (Musculoskeletal and connective tissue disorders) | 11 | 6
Cellulitis (Infections and infestations) | 5 | 3
GI Bleed (Gastrointestinal disorders) | 4 | 7
Myocardial infarction (Cardiac disorders) | 3 | 6
Bowel obstruction (Gastrointestinal disorders) | 8 | 1
Infection (Infections and infestations) | 6 | 9
Syncope/dizziness (Nervous system disorders) | 4 | 5
Misc. cardiac disorders (Cardiac disorders) | 17 | 26
Misc. GI disorders (Gastrointestinal disorders) | 8 | 13
Misc. ear and labyrinth disorders (Ear and labyrinth disorders) | 3 | 1
Misc. nervous system disorders (Nervous system disorders) | 8 | 2
Misc. psychiatric disorders (Psychiatric disorders) | 3 | 2
Misc. reproductive and breast disorders (Reproductive system and breast disorders) | 6 | 5
Misc. vascular disorders (Vascular disorders) | 8 | 11
Misc. renal and urinary disorders (Renal and urinary disorders) | 9 | 14
Misc. hepatobiliary disorders (Hepatobiliary disorders) | 5 | 4
Misc. metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 | 2
Misc. respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Misc. musculoskeletal disorders (Musculoskeletal and connective tissue disorders) | 8 | 4
Miscellaneous (General disorders) | 1 | 1
Misc. neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Injury (Injury, poisoning and procedural complications) | 5 | 4
Misc. endocrine disorders (Endocrine disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes